CLINICAL TRIAL: NCT03371082
Title: An Open Label, Randomized, Multicenter, Phase 3 Study to Compare the Immunogenicity, Efficacy and Safety of Gan & Lee Pharmaceuticals Insulin Glargine Injection to Lantus in Adult Subjects With Type 1 Diabetes Mellitus.
Brief Title: Gan & Lee Insulin Glargine Target Type (1) Evaluating Research
Acronym: GLITTER1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL-GLAT1-3001
Record Dates: First submitted 2017-11-20; First posted 2017-12-13 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Diabetes Type 1; Type 1; Basal; Insulin; Glargine; T1DM; Diabetes Mellitus; Insulin Dependent Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — gallium nitrate; Insulin Glargine

STUDY DESIGN:
Intervention Model Description: Subjects who meet the study eligibility criteria will be centrally randomized 1:1 in an open-label fashion to receive either Gan & Lee Insulin Glargine Injection or Lantus® for 26 weeks. Randomization will be stratified by country.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gan & Lee Insulin Glargine Injection (Experimental): Gan & Lee Insulin Glargine Injection for subcutaneous injection, 100 U/mL, in the integrated, disposable 3.0-mL pre-filled Gan & Lee injector pen. Subjects randomized to the Gan & Lee Insulin Glargine Injection group will participate in the study for 26 weeks.
  Interventions: Biological: Gan & Lee Insulin Glargine Injection
- Lantus® (Active Comparator): Lantus® (insulin glargine injection) solution for subcutaneous injection, 100 U/mL, in the SoloStar® 3.0 mL pre-filled insulin pen. Subjects randomized to the Lantus® group will participate for 26 weeks.
  Interventions: Biological: Lantus®

INTERVENTIONS:
Biological: Gan & Lee Insulin Glargine Injection — Route of administration: subcutaneous injection
  Arms: Gan & Lee Insulin Glargine Injection
Biological: Lantus® — Route of administration: subcutaneous injection
  Arms: Lantus®

SUMMARY:
Primary Objective:

•To evaluate equivalence of Gan & Lee Insulin Glargine Injection and Lantus® in terms of immunogenicity

Secondary Objective:

Immunogenicity:

• To evaluate the percentage of subjects with negative anti-insulin antibodies (AIAs) at baseline who develop confirmed positive AIA up to Week 26, the percentage of baseline in AIA titers between treatment groups, the percentage of subjects with confirmed positive AIA who develop any anti-insulin neutralizing antibodies up to visit Week 26, and percentage of subjects who develop confirmed positive AIA up to visit Week 26 of Gan & Lee Insulin Glargine Injection in comparison with that of Lantus®.

Safety:

•To evaluate the safety of Gan & Lee Insulin Glargine Injection in comparison with that of Lantus®.

Efficacy:

•To evaluate the efficacy of Gan & Lee Insulin Glargine Injection in comparison with that of Lantus®.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant, nonlactating female subjects between the ages of 18 and 75 years, inclusive.
2. Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with the ICH GCP Guideline E6 and all applicable regulations, before initiating any study-related procedures.
3. Ability to understand and fully comply with all study procedures and restrictions.
4. Subjects with a confirmed diagnosis of type 1 diabetes mellitus who have been on an approved basal and bolus insulin regimen for at least 6 months (the type or brand of insulin should not have changed in the 6 months before screening).
5. HbA1c ≤ 11.0%.
6. BMI ≥ 19 kg/m2 and ≤ 35 kg/m2.
7. Adherence to a prudent diet and exercise regimen recommended by the medical provider, and willingness to maintain these consistently for the duration of the study.
8. Concomitant medications are allowed, provided that no significant dosing changes are anticipated during the study (see the exclusion criteria below for specific prohibited concomitant medications); for concomitant thyroid medications, subjects must have been on a stable dosage for 90 days before screening.

Exclusion Criteria:

1. Participation in another clinical study or use of any study drug within 30 days before screening.
2. Previous use of a biosimilar insulin, either basal or bolus.
3. Diabetic ketoacidosis within a year before screening.
4. Brittle type 1 diabetes mellitus within the year before screening (e.g., multiple hospitalizations related to diabetes mellitus and/or severe hypoglycemia for which the subject required 3rd party assistance).
5. Any severe, delayed sequela of diabetes mellitus, e.g., worsening end-stage renal disease, advanced coronary artery disease, or myocardial infarction within the year before screening, or autonomic peristaltic problems, e.g., gastroparesis.
6. Anticipated change in insulin used during the study (change in dosage is allowed, but change in type or brand of insulin will result in the subject being withdrawn from the study).
7. Inadequately controlled thyroid disease, defined as a TSH or free T4 value > the upper limit of normal.
8. BMI < 19 kg/m2 or > 35 kg/m2.
9. Any clinically significant (in the opinion of the Investigator) hematology or chemistry test results at screening, including any liver function test > 3x the upper limit of normal (subjects with elevated bilirubin due to Gilbert syndrome are eligible to participate).
10. Documented history of anti-insulin antibodies.
11. Treatment with glucocorticosteroids, immunosuppressants, or cytostatic agents within 60 days before screening (newly-prescribed or high-dose corticosteroids are prohibited; chronically administered oral, inhaled, topical, or intra-articular corticosteroids at a stable dosage are allowed if no increase in dose is anticipated during the study; See Appendix 3 [Section 17.3] for a list of allowed and prohibited medications).
12. Current use of medication intended to cause weight loss or weight gain.
13. Alcohol or substance use disorder within the 2 years before screening.
14. Any previous or anticipated treatment with interferons.
15. Any history of malignant disease within 5 years before screening, except for adequately treated basal cell carcinoma.
16. Severe concomitant physical or psychiatric diseases or conditions
17. A history of a positive test result for HIV, hepatitis B, or hepatitis C; any subject who has a positive test result during the study may continue at the discretion of the Investigator.
18. Any history of pancreatitis or pancreatectomy.
19. Any diagnosis or condition that requires the subject to undergo procedures that could decrease antibodies in plasma or that would require treatment with immunosuppressant agents.
20. Any condition e.g., splenectomy, autoimmune disease, or rheumatologic disease, that could affect immunologic responses, could indicate an altered immune system, or could require treatment with a prohibited medication.
21. Any unresolved infection or a history of active infection within 30 days before screening other than mild or viral illness (as judged by the Investigator).
22. Any other disease or condition that in the opinion of the Investigator could confound the study results or limit the subject's ability to participate in the study or comply with follow-up procedures; or any other factor that would indicate a significant risk of loss to follow up.
23. Intolerance or history of hypersensitivity to insulin glargine or any excipient of IP.
24. Inability or unwillingness to wear the CGM sensor as required for the study, or to comply with the concomitant medication requirements in the FreeStyle Libre Pro Indications and Important Safety Information, during the CGM periods.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jia Lu, MD, PhD, Study Director — Gan & Lee Pharmaceuticals, USA; Elena A. Christofides, MD,FACE, Principal Investigator — Endocrinology Research Associates, Inc.
Locations (85):
- United States (50):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Valley Research, Fresno, California
  - The Rose Salter Medical Research Foundation, Newport Beach, California
  - California Medical Research Association, Northridge, California
  - Metabolic Institute of America, Tarzana, California
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Meridien Research, Bradenton, Florida
  - The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Homestead Associates in Research, Homestead, Florida
  - Central Florida Endocrine and Diabetes Consultants - Maitland, Maitland, Florida
  - Biotech Pharmaceutical Group, LLC, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Peninsula Research, Ormond Beach, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Sestron Clinical Research, Marietta, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Advanced Clinical Research - Idaho, Meridian, Idaho
  - Cedar Crosse Research Center, Chicago, Illinois
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Midwest CRC, Crystal Lake, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Physicians East - Greenville, Greenville, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Endocrinology Reserach Associates, Inc., Columbus, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - ClinSearch - Clinical Research Specialists, Chattanooga, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - Texas Diabetes & Endocrinology - Central Austin, Austin, Texas
  - Texas Diabetes & Endocrinology - South Austin, Austin, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Texas Diabetes & Endocrinology - Round Rock, Round Rock, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Northeast Clinical Research of San Antonio, Schertz, Texas
  - Radiant Research, Murray, Utah
  - Advanced Research Institute, Ogden, Utah
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Burke Internal Medicine & Research, Burke, Virginia
  - Stonesifer Clinical Research, Federal Way, Washington
  - Rainier Clinical Research Center, Inc., Renton, Washington
  - MultiCare Health System Institute for Research & Innovation, Tacoma, Washington
- Czechia (7):
  - Diabetologie České Budějovice s.r.o, České Budějovice, Jihočeský kraj
  - Krajská zdravotní, a.s., Masarykova nemocnice v Ústí nad Labem, Ústí nad Labem, Severoceský KRAJ
  - Diahaza s.r.o., Holešov
  - StefaMed, Hradec Králové
  - Diabetologie MUDr. Tomáš Edelsberger, Krnov
  - PreventaMed, Olomouc
  - Genom s.r.o, Ostrava
- Germany (6):
  - Studienzentrum Aschaffenburg, Aschaffenburg, Bavaria
  - Diabetes-falkensee.de, Falkensee, Brandenburg
  - Gemeinschaftspraxis Diabeteszentrum Dortmund, Dortmund, North Rhine-Westphalia
  - Diabetes Schwerpunktpraxis, Gemeinschaftspraxis Alain Barakat und Helene Willems, Duisburg, North Rhine-Westphalia
  - Diabetologische Schwerpunktpraxis Pirna, Pirna, Saxony
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
- Hungary (7):
  - CRU Hungary Egészségügyi és Szolgáltató Kft., Miskolc, Borsod-Abauj Zemplen county
  - Lausmed Egeszsegugyi es Szolgaltato Kft., Baja, Bács-Kiskun county
  - Markhot Ferenc Oktatókórház és Rendelointézet, Eger, Heves County
  - Zala County Hospital, Zalaegerszeg, Zala County
  - Betegapolo-Irgalmasrend Budai Irgalmasrendi Kórház, Diabetológiai Ambulancia, Budapest
  - Synexus Magyarország, Budapest
  - Semmelweis Egyetem II. Sz. Belgyógyászati Klinika, Budapest
- Poland (7):
  - Praktyka Lekarska Ewa Krzyzagórska, Poznan, Greater Poland Voivodeship
  - Pratia MCM Kraków, Krakow, Lesser Poland Voivodeship
  - NZOZ Medyczne Centrum Diabetologiczno-Endokrynologiczno-Metaboliczne "Diab-Endo-Met", Krakow, Lesser Poland Voivodeship
  - KO-MED Centra Kliniczne Lublin - Królewska, Lublin, Lublin Voivodeship
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administracji w Warszawie, Warsaw, Masovian Voivodeship
  - Centrum Badań Klinicznych PI-House, Gdansk, Pomeranian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Gdanska Poradnia Cukrzycowa, Gdansk, Pomeranian Voivodeship
- Spain (8):
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona, Gerona
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, LA Coruna
  - Centro de Especialidades San Jose Obrero. Hospital Universitario Virgen de la Victoria, Málaga, Malaga
  - Complejo Hospitalario Universitario La Coruña, A Coruña
  - Hospital Universitario Ramón Y Cajal, Madrid
  - Nuevas Tecnologías en Diabetes y Endocrinología, Seville
  - Hospital Universitario Nuestra Señora de Valme, Seville
  - Consorci Hospital General Universitari de València, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Reviewed and approved by each IRB.
Period: Overall Study
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Started | 287 | 289
Completed | 258 | 255
Not Completed | 29 | 34

BASELINE CHARACTERISTICS:
Population: All Subjects Assigned randomly to treatment (full analysis set).
Groups:
- Total: Total of all reporting groups
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus® | Total
Number analyzed (Participants) | 287 | 289 | 576
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 256 | 252 | 508
  >=65 years | 31 | 37 | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.7 (13.96) | 46.7 (14.46) | 46.2 (14.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 112 | 215
  Male | 184 | 177 | 361
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 16 | 39
  Not Hispanic or Latino | 259 | 272 | 531
  Unknown or Not Reported | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 13 | 14 | 27
  White | 262 | 265 | 527
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Hungary | 20 | 21 | 41
  United States | 151 | 150 | 301
  Czechia | 24 | 25 | 49
  Poland | 37 | 37 | 74
  Germany | 29 | 28 | 57
  Spain | 26 | 28 | 54
Anti-Insulin Antibodies (AIA) [Count of Participants; unit: Participants]
  Negative | 236 | 239 | 475
  Positive | 49 | 48 | 97
  Nonreportable | 0 | 2 | 2
  Missing | 2 | 0 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 27.01 (3.875) | 27.11 (4.237) | 27.06 (4.058)
Duration of Diabetes [Mean (Standard Deviation); unit: Years] | 20.2 (13.88) | 21.7 (13.95) | 21.0 (13.92)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: HbA1c (%)] | 8.11 (1.229) | 8.08 (1.267) | 8.10 (1.247)
Anti-Insulin Neutralizing Antibodies (NAbs) [Count of Participants; unit: Participants]
  Negative | 44 | 38 | 82
  Positive | 6 | 9 | 15
  Missing | 1 | 1 | 2
  Not Tested | 236 | 241 | 477
Thyroid Disease [Number; unit: Participants]
  Absence | 243 | 210 | 453
  Presence | 44 | 79 | 123
  Hypothyroidism | 32 | 52 | 84
  Hyperthyroidism | 1 | 5 | 6
  Structural abnormality | 5 | 4 | 9
  Thyroid Cancer | 0 | 0 | 0
  Other | 6 | 18 | 24
Weight [Mean (Standard Deviation); unit: kg] | 80.901 (13.4277) | 81.548 (16.3993) | 81.226 (14.9829)

OUTCOME MEASURES:

1. Primary Outcome: Treatment-induced Anti-Insulin Antibody (TI-AIA)
Description: TI-AIA is the Composite of Newly Confirmed Positive AIA or Important-Increase in AIA titer
Time Frame: Assessed up to Week 26
Population: The Safety Analysis Set (SS) was comprised of all subjects whose treatment assignment was randomly assigned who received any of the study treatment, even a partial dose, and had non-missing values.
Measure: Mean (Standard Deviation); unit: Titers
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 287 | 289
Titers | 4.8 (88.88) | 42.5 (332.90)
Statistical Analysis 1: Comparison: Gan & Lee Insulin Glargine Injection vs Lantus®; This is a two-arm study; Test type: Equivalence — The limits of the lower and upper equivalence margin were -11.3 and 11.3, respectively; Risk Difference (RD) = 0.6, 90% CI 2-sided [-5.4 to 6.5], Standard Error of Mean 3.63 — The asymptotic standard error was planned and is reported above

2. Secondary Outcome: Glycosylated Hemoglobin HbA1c
Description: The change between baseline (CFB) in HbA1c and at 26 weeks
Time Frame: Assessed up to Week 26
Population: The Full Analysis Set (FAS) was comprised of all subjects whose treatment assignment was randomly assigned with non-missing baseline values.
Measure: Least Squares Mean (Standard Error); unit: Percent of total hemoglobin
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 287 | 289
Percent of total hemoglobin | -0.08 (0.072) | 0.00 (0.061)

3. Secondary Outcome: Number of Subjects in Each Treatment Group With Negative AIA at Baseline Who Develop Confirmed Positive AIA After Baseline
Description: The number of subjects in each treatment group with negative AIA at baseline who develop confirmed positive AIA after baseline and up to visit Week 26.
Time Frame: Assessed up to Week 26
Population: Subset of subjects whose baseline AIA was negative (n=475).
Measure: Count of Participants; unit: Participants
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 236 | 239
Participants | 63 | 59

4. Secondary Outcome: Number of Subjects in Each Treatment Group With Confirmed Positive AIA at Baseline and at Least a 4-fold Increase in Titers After Baseline.
Description: The number of subjects in each treatment group with confirmed positive AIA at baseline and at least a 4-fold increase in titers after baseline and up to 26 weeks.
Time Frame: Up to Week 26
Population: Subset of subjects whose baseline AIA was confirmed positive (n=97).
Measure: Count of Participants; unit: Participants
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 49 | 48
Participants | 11 | 14

5. Secondary Outcome: Mean Change From Baseline in Each Treatment Group in AIA Titers After Baseline
Description: The mean change from baseline in each treatment group in AIA titers after baseline and up to visit Week 26.
Time Frame: Assessed up to Week 26
Population: Subjects with Confirmed Positive Anti-Insulin Antibodies at Baseline with non-missing AIA titer values.
Measure: Mean (Standard Deviation); unit: Titers
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 29 | 30
Titers | 4.8 (88.88) | -42.5 (332.90)

6. Secondary Outcome: Number of Subjects With Confirmed Positive AIA After Baseline Who Develop Any Anti-insulin Neutralizing Antibodies After Baseline.
Description: The number of subjects in each treatment group with confirmed positive AIA after baseline and up to visit Week 26 who develop any anti-insulin neutralizing antibodies after baseline and up to visit Week 26.
Time Frame: Up to Week 26
Population: Safety Analysis Set - Subjects with Confirmed Positive AIA after Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 54 | 60
Participants | 13 | 16

7. Secondary Outcome: Number of Subjects With Confirmed Positive AIA After Baseline.
Description: The number of subjects in each treatment group with confirmed positive AIA after baseline and up to visit Week 26.
Time Frame: Up to Week 26
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 287 | 289
Participants | 102 | 103

8. Secondary Outcome: Postbaseline FBG Control
Description: The number of subjects who achieve an FBG test result of ≤ 6.0 mmol/L at visit Week 26.
Time Frame: Up to Week 26
Population: FBG control (FBG ≤ 6.0 mmol/L).
Measure: Count of Participants; unit: Participants
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 287 | 289
Participants
  Lack of Postbaseline FBG control | 248 | 247
  Sufficient Postbaseline FBG control | 39 | 42

9. Secondary Outcome: HbA1c Control.
Description: The number of subjects who achieve a HbA1c of < 7.0% at visit Week 26.
Time Frame: Up to Week 26
Population: HbA1c control (HbA1c < 7.0%).
Measure: Count of Participants; unit: Participants
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 287 | 289
Participants
  Lack of Postbaseline HbA1c Control | 241 | 245
  Sufficient Postbaseline HbA1c Control | 46 | 44

ADVERSE EVENTS:
Time Frame: 26-weeks
Description: All untoward events, All-Cause Mortality, Serious, or Any Other (non-serious) Adverse Events were collected by regular investigator assessment and participants self-report, monitored, assessed, coded, and summarized.
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
All-Cause Mortality (participants affected / at risk) | 0/287 | 1/289
Serious Adverse Events (participants affected / at risk) | 10/287 | 14/289
Other Adverse Events (participants affected / at risk) | 160/287 | 161/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gan & Lee Insulin Glargine Injection (N=287) | Lantus® (N=289)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (20) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Appendicitis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Benign neoplasm of spinal cord (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Vascular disorders) | 0 (0) | 1 (1)
Cough (General disorders) | 0 (0) | 1 (1)
Craniocerebral injury (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Endocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Inguinal Hernia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower limb fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peripheral ischemia (Vascular disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Post procedural infection (General disorders) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rib fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Septic shock (General disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Thrombosis (General disorders) | 1 (1) | 0 (0)
Tibia fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gan & Lee Insulin Glargine Injection (N=287) | Lantus® (N=289)
Hypoglycemia (Metabolism and nutrition disorders) | 158 (3476) | 161 (2936)
Weight increase (Investigations) | 3 (3) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4) | 1 (3)
Blood creatine phosphokinase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Contusion (General disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Face oedema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Foot Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Herpes zoster (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT03371082/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT03371082/SAP_001.pdf
  • Informed Consent Form (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT03371082/ICF_002.pdf